CLINICAL TRIAL: NCT04246866
Title: A Phase 1, Multicenter, Open-label, Single-dose, Dose-escalation Study in Patients With Geographic Atrophy (GA) Secondary to Dry Age-related Macular Degeneration (AMD) to Evaluate the Safety, Tolerability, Pharmacodynamics, and Immunogenicity of Intravitreal Injections of GEM103
Brief Title: First in Human Study to Evaluate the Safety and Tolerability of GEM103 in Geographic Atrophy Secondary to Dry Age Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gemini Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEM-CL-10301
Record Dates: First submitted 2020-01-06; First posted 2020-01-29 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Dry Age-related Macular Degeneration; Geographic Atrophy; Macular Degeneration; Retinal Disease; Retinal Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration; Retinal Diseases; Retinal Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose 1 (Experimental): A single dose of GEM103 will be administered via intravitreal injection. This arm will be the lowest dose of GEM103
  Interventions: Biological: GEM103
- Dose 2 (Experimental): A single dose of GEM103 will be administered via intravitreal injection. This arm will be the medium dose of GEM103
  Interventions: Biological: GEM103
- Dose 3 (Experimental): A single dose of GEM103 will be administered via intravitreal injection. This arm will be a higher dose of GEM103
  Interventions: Biological: GEM103
- Dose 4 (Experimental): A single dose of GEM103 will be administered via intravitreal injection. This arm will be the highest (extension) dose of GEM103
  Interventions: Biological: GEM103

INTERVENTIONS:
Biological: GEM103 — GEM103

SUMMARY:
The study is designed to identify the maximum tolerated dose (MTD) for intravitreal (IVT) administration of GEM103 in subjects with geographic atrophy (GA) secondary to dry AMD. Safety and tolerability of a single dose of GEM103 will be assessed based on the occurrence of dose-limiting toxicities (DLTs). Each subject will be followed for safety, pharmacokinetic (PK), clinical, and biomarker evaluations. Three escalating dose cohorts are planned.

DETAILED DESCRIPTION:
This is a Phase 1, multicenter, open-label, single-dose, dose-escalation study in subjects with GA secondary to dry AMD to investigate the safety, tolerability, pharmacodynamics (PD), and immunogenicity of IVT injections of GEM103 to a single eye.

The study is designed to identify the MTD for IVT administration of GEM103. Safety and tolerability of a single dose of GEM103 will be assessed based on the occurrence of DLTs. Three escalating dose cohorts are planned.

Subjects will undergo clinical and ophthalmic assessments for inclusion eligibility into the study. Enrolled subjects will receive GEM103 and be followed for safety, PK, clinical, and biomarker evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. At least 50 years old at the time of signed informed consent
2. Able to cooperate sufficiently for adequate ophthalmic visual function testing and anatomic assessment and provide informed consent prior to initiation of any study procedure
3. Best corrected visual acuity (BCVA) in study eye between 5-45 letters
4. Confirmed diagnosis of central GA in the study eye and eligible total GA lesion size

Exclusion Criteria:

1. Presence of the following ocular conditions - in the study eye:

   * Exudative AMD or choroidal neovascularization (CNV)
   * Any ocular disease or condition that could impact the subject's ability to participate in the study or be a contraindication to IVT injection
   * Any intraocular surgery (with the exception of intraocular lens replacement surgery more than 3 months prior to consent)
2. Presence of any of the following ocular conditions - in either eye:

   * History of herpetic infection
   * Ongoing treatment with antiangiogenic therapies in the fellow eye or completed treatment in the study eye
3. Any prior or ongoing medical condition (e.g. ocular other than dry AMD, systemic, psychiatric) or clinically significant screening laboratory value that may present a safety risk, interfere with study compliance, interfere with consistent study follow-up, or confound data interpretation throughout the longitudinal follow-up period
4. Female subjects must not be pregnant or lactating
5. Current use of medications known to be toxic to the lens, retina, or optic nerve

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2020-10-21 (Actual); Study Completion 2020-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of AEs/SAEs following drug administration | Up to 8 Weeks

SECONDARY OUTCOMES:
GEM103 concentrations in ocular fluids | Up to 8 Weeks
Changes in complement factor levels compared to baseline after drug administration | Up to 8 Weeks

OTHER OUTCOMES:
Change from baseline in aqueous humor biomarker levels (in ng/mL) of complement factors | Up to 8 Weeks
Change from baseline in clinical assessments including BCVA and LLVA scores as assessed by ETDRS Visual Acuity Score in number of letters | Up to 8 Weeks
Change from baseline in clinical assessments including area of GA in mm2 as assessed by fundus imaging | Up to 8 Weeks
Change in concentration of GEM103 in blood samples | Up to 8 Weeks

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Associated Retina Consultants, Phoenix, Arizona
  - Retinal Consultants of Arizona, Phoenix, Arizona
  - California Retina Consultants, Bakersfield, California
  - Retina Vitreous Associates, Beverly Hills, California
  - California Retina Consultants, Oxnard, California
  - California Retina Consultants, Santa Barbara, California
  - California Retina Consultants, Santa Maria, California
  - Southeast Retina Center, Augusta, Georgia
  - Midwest Eye Institute, Indianapolis, Indiana
  - Pepose Vision Institute, Chesterfield, Missouri
  - Sierra Eye Associates, Reno, Nevada
  - Western Carolina Retinal Associates, Asheville, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khanani AM, Maturi RK, Bagheri N, Bakall B, Boyer DS, Couvillion SS, Dhoot DS, Holekamp NM, Jamal KN, Marcus DM, Pieramici D, Aziz AA, Patki KC, Bridges WZ Jr, Barone SB. A Phase I, Single Ascending Dose Study of GEM103 (Recombinant Human Complement Factor H) in Patients with Geographic Atrophy. Ophthalmol Sci. 2022 Apr 11;2(2):100154. doi: 10.1016/j.xops.2022.100154. eCollection 2022 Jun. PMID 36249705